CLINICAL TRIAL: NCT00039780
Title: BNP7787 vs. Placebo for Prevention of Paclitaxel Neurotoxicity: A Double-Blind Multicenter Randomized Phase 3 Trial in Patients With Metastatic Breast Cancer
Brief Title: Evaluation of BNP7787 for the Prevention of Neurotoxicity in Metastatic Breast Cancer Patients Receiving Weekly Paclitaxel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNumerik Pharmaceuticals, Inc. (Industry)
Collaborators: Lantern Pharma Inc. became Sponsor of Tavocept (BNP7787) IND 051014 as of March 26, 2019. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMS30203R
Record Dates: First submitted 2002-06-10; First posted 2002-06-13 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Breast Neoplasms; Breast Diseases; Metastases, Neoplasm
Keywords: Breast; Cancer; Metastatic; Paclitaxel; Peripheral; Taxol; Neuropathy; Neurotoxicity; Paresthesias; Weekly; BNP7787; 7787; Tavocept; Prevention
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasm Metastasis; Neoplasms; Neurotoxicity Syndromes; Paresthesia | interventions — 2,2'-dithiodiethanesulfonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Tavocept (BNP7787)
  Interventions: Drug: BNP7787
- 2 (Placebo Comparator): 0.9% Sodium Chloride Soln.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BNP7787 — The treatment regimen administered in this study is a single IV doxe of paclitaxel (80 mg/m2) +/- Herceptin given over 1 hour and either BNP7787 (18.4 g/m2) or placebo given over 45 minutes each week. One treatment cycle = 8 weeks.
  Other Names: BNP7787 also known as Tavocept
  Arms: 1
Drug: Placebo — The treatment regimen administered in this study is a single IV doxe of paclitaxel (80 mg/m2) +/- Herceptin given over 1 hour and either BNP7787 (18.4 g/m2) or placebo given over 45 minutes each week. One treatment cycle = 8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether BNP7787 is effective in preventing or reducing neurotoxicity (nerve damage) caused by paclitaxel (Taxol®).

DETAILED DESCRIPTION:
Chemotherapy induced toxicities are common and serious problems for many patients who receive treatment for cancer. Chemotherapy induced toxicities can adversely impact the quality of life and the ability of patients to continue treatment for their cancer. One such toxicity associated with the use of paclitaxel (Taxol®) is peripheral neurotoxicity.

Paclitaxel is an active drug in the treatment of metastatic breast cancer as first-line treatment and in patients with recurrent or refractory disease, including patients who have failed to respond to previous anthracycline therapy. Recent studies with paclitaxel using a weekly schedule of administration have demonstrated higher tumor response rates and disease free survival accompanied by a shift in the frequency of certain toxicities, increased dose intensity and a potential means to improve the treatment schedule of paclitaxel for improved patient benefit.

Paclitaxel induced neurotoxicity remains an important problem that limits the ability to improve the schedule of administration of this drug. To date, there is no effective or FDA approved therapy to prevent the development of or reduce the frequency or severity of paclitaxel-induced neurotoxicity.

BNP7787 is an investigational new drug that is undergoing development for chemoprotection of platinum and taxane associated common clinical toxicities, particularly the prevention of chemotherapy-induced neurotoxicity.

In this Phase 3 clinical trial the safety and effectiveness of BNP7787 in preventing or mitigating the frequency, severity, worsening of grade, time to onset, duration and discontinuation of therapy due to paclitaxel-induced neurotoxicity will be assessed in patients with metastatic breast cancer.

ELIGIBILITY:
INCLUSION CRITERIA

Histologically or cytologically documented metastatic breast cancer

Measurable disease

Performance Status; ECOG 0-2

More than 2 weeks since prior radiation therapy

14 days or more since prior therapy and recovered from all side effects

For patients who progress while receiving hormonal therapy alone, the patient may be enrolled on study as soon as they have recovered from all side effects of the hormonal therapy

Clinical laboratory values must meet the following:

* Granulocytes greater than or equal to 1,500/mm(3)
* Platelets greater than or equal to 100,000/mm(3)
* Hemoglobin greater than or equal to 9 g/dL
* SGOT less than 2.0 x ULN
* Bilirubin less than or equal to 1.5 mg/dL
* Creatinine less than or equal to 1.6 mg/dL
* Calcium less than the ULN

EXCLUSION CRITERIA

Current CNS metastases or history of CNS metastases

History of diabetes (Type I or Type II)

Previous or concurrent malignancy except:

* inactive non-melanoma skin cancer
* in situ carcinoma of the cervix
* or other cancer if the patient has been disease-free for more than 5 years

Pregnant or lactating women

History of recent myocardial infarction, stroke, or uncontrolled CHF, epilepsy, or hypertension

Patients currently receiving Neurontin® (gabapentin), glutamine supplements, Elavil® (amitriptyline), Dilantin®, Tegretol®, tricyclic antidepressants or other similar medications during the study period

Alternative medications including megadose vitamins, herbal preparations, tonics, extracts, etc. are not allowed during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2001-09; Primary Completion 2006-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
1)Incidence of PNQ Grade D or Grade E neurosensory symptoms (Item 1 of the PNQ) with duration of at least 4 weks; 2) Objective tumor response rate | baseline to disease progression or discontinuation from study

SECONDARY OUTCOMES:
Incidence of Dose Modifications, Treatment Delays and Treatment Discontinuations due to Neurotoxicity | baseline to end of treatment
Time-to-onset of clinically important neurotoxicity | randomization to date of first occurrence of clinically important neurotoxicity
Incidence of Neurosensory and Neuromotor Functional Impairment | baseline through end of treatment
Progression Free Survival | Randomization to disease progression or death due to any cause